CLINICAL TRIAL: NCT02981303
Title: A Multicenter, Open-label, Phase 2 Study of Imprime PGG and Pembrolizumab in Subjects With Advanced Melanoma Failing Front-line Treatment With Checkpoint Inhibitors (CPI) or TNBC Failing Front-line Chemotherapy for Metastatic Disease
Brief Title: Study of Imprime PGG and Pembrolizumab in Advanced Melanoma and Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HiberCell, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-CL-PGG-MEL/BCA-1621/MK3475
Record Dates: First submitted 2016-11-22; First posted 2016-12-05 (Estimated); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Advanced Melanoma; Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melanoma (Experimental): Imprime PGG + Pembrolizumab
  Interventions: Biological: Imprime PGG; Drug: Pembrolizumab
- Triple Negative Breast Cancer (Experimental): Imprime PGG + Pembrolizumab
  Interventions: Biological: Imprime PGG; Drug: Pembrolizumab

INTERVENTIONS:
Biological: Imprime PGG — Imprime PGG is a soluble, β-1,3/1,6 glucan isolated from the cell wall of a proprietary Saccharomyces cerevisiae yeast strain. Imprime PGG acts as a Pathogen-Associated Molecular Pattern (PAMP). Imprime will be administered at a dose of 4 mg/kg IV over a 2-hour infusion time on Days 1, 8 and 15 of each 3-week treatment cycle.
  Other Names: Imprime
Drug: Pembrolizumab — Pembrolizumab is a humanized monoclonal antibody against the programmed death receptor-1 protein. Pembrolizumab will be given at a fixed dose of 200 mg IV over 30 minutes on Day 1 of each 3-week treatment cycle after the Imprime infusion.
  Other Names: Keytruda

SUMMARY:
Objective: To determine the Overall Response Rate (ORR) to Imprime PGG + pembrolizumab in subjects with advanced melanoma or metastatic TNBC

Safety: To characterize the safety of Imprime PGG + pembrolizumab given in combination

Hypothesis: Restore (for melanoma) or enhance (for TNBC) sensitivity to checkpoint inhibitors (CPI) by appropriate and effective stimulation of the subject's innate and adaptive immune systems in those subjects who have failed 1st line therapy

The study will incorporate Simon's optimal 2-stage design with sample size fixed at 12 subjects each in Stage 1 for advanced melanoma and for Triple Negative Breast Cancer (TNBC) subjects. The safety criterion of ≤ 4 (or ≤ 33%) subjects with Grade 3/4 adverse events in Cycle 1 within either tumor type must be met in order to proceed to Stage 2. The starting dose is 4 mg/kg for Imprime PGG. In the event there are a total of > 4 (or > 33%) of subjects with Grade 3/4 adverse events in Cycle 1, the dose of Imprime PGG will be reduced to 2 mg/kg, and Stage 1 will be repeated at a dose of 2 mg/kg with an additional cohort of n=12 subjects. For the dose that meets the safety criterion in Stage 1, at least 1 response in melanoma subjects and 2 responses in TNBC subjects amongst the 12 subjects within each tumor type must be observed in order to proceed to Stage 2.

Stage 2 will enroll an additional 17 subjects with melanoma, and 30 subjects with TNBC. For the dose that meets the Stage 1 safety criterion, success will be declared if at least 4 amongst the total of up to 29 subjects with melanoma, and 13 amongst the total of up to 42 subjects with TNBC achieve an objective response.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed an informed document prior to any study-specific procedures or treatment
2. Be ≥ 18 years of age at time of consent
3. For Melanoma Subjects: Have histologically or cytologically confirmed diagnosis of unresectable Stage III or metastatic (Stage IV) melanoma not amenable to local therapy, and irrespective of PD-L1 status
4. For TNBC Subjects: Have histologically or cytologically confirmed diagnosis of metastatic (Stage IV) TNBC, and irrespective of PD-L1 status. TNBC is defined as negative immunohistochemistry (IHC) assays for Estrogen Receptor (ER), and Progesterone Receptor (PR), and HER2 negative (IHC 0 or 1+, or 2+ by IHC confirmed negative by FISH)
5. Have documented objective radiographic or clinical disease progression after PD-1/PD-L1 +/- anti-CTLA-4 inhibitor therapy (melanoma) or after at least 1 line of chemotherapy for metastatic disease (TNBC)
6. Have resolution of all previous treatment-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy (less than or equal to Grade 2) or alopecia. If subject received major surgery or radiation therapy of > 30 Gy, must have recovered from the toxicity and/or complications from the intervention.
7. Have at least one radiologically measurable lesion as per RECIST v1.1 defined as a lesion that is at least 10 mm in longest diameter or lymph node that is at least 15 mm in short axis imaged by CT scan or MRI and obtained by imaging within 28 days prior to start of study treatment. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. Have peripheral blood levels of IgG anti-β-glucan antibody (ABA) of ≥ 20 mcg/mL as determined by an ELISA test within 28 days prior to start of study treatment
9. Be willing to consider providing fresh tissue for biomarker analysis, and, based on the adequacy of the tissue sample quality, for assessment of biomarker status. Repeat samples may be required if adequate tissue is not provided. Newly obtained biopsy specimens are preferred to archived samples and formalin-fixed, paraffin-embedded block specimens are preferred to slides.

   Note: Information on 1 tumor biopsy sample is mandatory and is as follows: (1) To determine eligibility, historical (diagnostic) tumor biopsy official pathology report +/- an archival sample. Additional biopsy samples, preferably obtained from the same localized region, are highly desirable when feasible at the following time points: (2) Sample before the first dose of study treatment, (3) Sample after completion of Cycle 2 but before the start of Cycle 3 dosing, and (4) Sample either at the time of response or at the End of Study Visit (if no response).
10. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (see Appendix 14.3)
11. Have life expectancy of 3 months or greater as determined by the treating physician
12. Have adequate organ function (all screening labs should be performed within 15 days prior to treatment initiation):

    1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN
    2. Aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
    3. Alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
13. Have adequate renal function as defined by the following criteria:

    Creatinine ≤ 1.5 x ULN and CrCl ≥ 30 ml/min per Cockcroft Gault formula:
14. Have adequate hematologic function, defined as meeting all of the following criteria:

    1. Hemoglobin ≥ 9 g/dL (uncorrected by RBC transfusion)
    2. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
    3. Platelet count ≥ 100 × 109/L
15. Have adequate coagulation functioning within 15 days prior to start of study treatment, defined by either of the following criteria:

    1. INR < 1.5 × ULN
    2. OR for subjects receiving warfarin or low molecular weight heparin (LMWH), the subjects must, in the Investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for these subjects may exceed 1.5 × ULN if that is the goal of anticoagulant therapy.
    3. Activated Partial Thromboplastin Time (aPTT) < 1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
16. Female subjects of childbearing potential as defined in Section 5.7.2 must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
17. If of childbearing potential as defined in Section 5.7.2, must be willing to use an adequate method of contraception (see Section 5.7.2) from the first dose of study medication through 120 days after the last dose of study medication
18. Be willing and have the ability to comply with scheduled visits (including geographical proximity), treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

1. Has disease that is suitable for local therapy administered with curative intent
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
3. Has a diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
4. Has known history of active tuberculosis
5. Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
6. Has known active Hepatitis B (eg, HBsAg reactive) or Hepatitis C (eg, HCV RNA [qualitative] is detected
7. Has a history of clinically severe autoimmune disease, or history of organ transplant
8. Has a history of ocular melanoma
9. Has known hypersensitivity to baker's yeast
10. Had previous exposure to Betafectin® or Imprime PGG
11. Has hypersensitivity to pembrolizumab or any of its excipients
12. Had a prior anti-cancer monoclonal antibody (except immune CPI in the case of melanoma subjects) within 30 days prior to start of study treatment, or failure to recover to CTCAE Grade 1 or better from the adverse events of prior therapies
13. Had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Study Day 1 or who has not recovered from adverse events due to a previously administered agent or major surgery
14. Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF, or recombinant erythropoietin) within 4 weeks prior to Study Day 1
15. Has known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
16. Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
17. Has active autoimmune disease requiring systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
18. Has evidence of (non-infectious) pneumonitis that required steroids or current pneumonitis
19. Has a history of interstitial lung disease
20. Has an active infection requiring systemic therapy
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator
22. Has a clinically significant cardiovascular disease such as unstable angina, myocardial infarction, or acute coronary syndrome within ≤180 days prior to start of study treatment, symptomatic or uncontrolled arrhythmia, congestive heart failure, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
23. Has a known psychiatric or substance abuse disorder(s) that would interfere with informed consent or cooperation with the requirements of the trial
24. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
25. With TNBC has received prior therapy with an anti-PD-1, anti-PD-L1, anti-CTLA-4, or anti-PD-L2 agent
26. Has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Graff, PhD, Study Director — HiberCell, Inc.
Locations (10):
- United States (10):
  - Arizona Center for Cancer Care, Avondale, Arizona
  - John Wayne Cancer Institute, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Sarah Cannon Research Institute, Denver, Colorado
  - University Cancer and Blood Center, Athens, Georgia
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Thomas Jefferson University Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Millennium Oncology, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alison Stopeck, Michele Anne Gargano, Nick Niles, Blaine Rathmann, Michael Jon Chisamore, Nandita Bose, and Jose Luis Iglesias. A multicenter, open-label, phase 2 study of odetiglucan (IMPRIME PGG) and pembrolizumab in patients with metastatic breast cancer (mBCA) who have progressed through prior hormonal therapy. Journal of Clinical Oncology. 2022; Volume 40, Number 16_suppl. https://doi.org/10.1200/JCO.2022.40.16_suppl.TPS1115
- [Background] Chan ASH, Kangas TO, Qiu X, Uhlik MT, Fulton RB, Ottoson NR, Gorden KB, Yokoyama Y, Danielson ME, Jevne TM, Michel KS, Graff JR, Bose N. Imprime PGG Enhances Anti-Tumor Effects of Tumor-Targeting, Anti-Angiogenic, and Immune Checkpoint Inhibitor Antibodies. Front Oncol. 2022 May 26;12:869078. doi: 10.3389/fonc.2022.869078. eCollection 2022. PMID 35692755
- [Result] Steven O'Day, Virginia F. Borges, Bartosz Chmielowski, Ruta D. Rao, Maysa M. Abu-Khalaf, Alison Stopeck, Petros Nikolinakos, Melinda L. Telli, Bin Xie, Montaser F. Shaheen, Paulette Mattson, Michele Anne Gargano, Joanna Cox, Vassiliki Karantza, Michael Jon Chisamore, Bruno Osterwalder, Nandita Bose, Mark T. Uhlik, and Jeremy Graff. An open label, multicenter phase II study combining imprime PGG (PGG) with pembrolizumab (P) in previously treated metastatic triple-negative breast cancer (mTNBC). Journal of Clinical Oncology. 2019; Volume 37, Number 15_suppl. https://doi.org/10.1200/JCO.2019.37.15_suppl.2550
- [Result] Uhlik M, et al. Response and clinical benefit assessment of the combination of the Dectin-1 agonist Imprime PGG and anti-PD-1 Pembrolizumab in chemotherapy-resistant metastatic triple negative breast cancer. San Antonio Breast Cancer Symposium. 2019. PD-02.
- [Result] Breast Cancer Plenary Session: O'Day S, et al. A phase 2 trial of pembrolizumab and a novel innate immune activator, Imprime PGG, in metastatic triple negative breast cancer. AACR 2020. (#10531)
- [Result] Late Breaking Abstract: Chan ASH, et al. Clinical benefit evident with early immunopharmacodynamic responses in prior-checkpoint failed metastatic melanoma patients treated with Imprime PGG and Pembrolizumab. SITC 2019. (#P862)
- [Derived] Stopeck AT, Abu-Khalaf M, Borges V, Chmielowski B, Rao R, Xie B, Dudek AZ, Mina L, O'Shaughnessy J, Chisamore M, Mattson P, Gargano M, Cox J, Osterwalder B, Drees J, Harrison B, Chan ASH, Qiu X, Ottoson N, Bose N, Uhlik M, Graff J, Iglesias J. Phase 2 trial of imprime and pembrolizumab immunotherapy in metastatic triple negative breast cancer patients who have progressed beyond first line chemotherapy. J Immunol. 2025 Jul 1;214(7):1529-1538. doi: 10.1093/jimmun/vkaf079. PMID 40338159

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included arms with independent Simon 2-stage designs with 29 planned for the melanoma arm (12 subjects in Stage 1 and 17 subjects in Stage 2) and 41 planned for the TNBC arm (12 patients in Stage 1 and 29 patients in Stage 2) for a total of 60 subjects enrolled competitively across US clinical sites.
Groups:
- Melanoma: 4 mg/kg Imprime PGG + 200 mg IV every 3 weeks (Q3W) pembrolizumab in subjects with advanced melanoma
  Pembrolizumab: Pembrolizumab is a humanized monoclonal antibody against the programmed death receptor-1 protein. Pembrolizumab will be given at a fixed dose of 200 mg IV over 30 minutes on Day 1 of each 3-week treatment cycle after the Imprime infusion.
- Triple Negative Breast Cancer: 4 mg/kg Imprime PGG + 200 mg IV every 3 weeks (Q3W) pembrolizumab in subjects with metastatic TNBC
  Pembrolizumab: Pembrolizumab is a humanized monoclonal antibody against the programmed death receptor-1 protein. Pembrolizumab will be given at a fixed dose of 200 mg IV over 30 minutes on Day 1 of each 3-week treatment cycle after the Imprime infusion.
Period: Overall Study
Arm/Group | Melanoma | Triple Negative Breast Cancer
Started | 20 | 44
Completed | 2 | 2
Not Completed | 18 | 42
Not completed — Progressive Disease | 17 | 37
Not completed — Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects screened for the study who received at least one dose of study drug (primary population for baseline characteristics and safety analyses and secondary population for efficacy analyses).
Groups:
- Arm 1/ Melanoma: Arm 1: 4 mg/kg Imprime PGG + 200 mg IV every 3 weeks (Q3W) pembrolizumab in subjects with advanced melanoma
- Arm 2/ TNBC: Arm 2: 4 mg/kg Imprime PGG + 200 mg IV every 3 weeks (Q3W) pembrolizumab in subjects with metastatic TNBC
- Total: Total of all reporting groups
Arm/Group | Arm 1/ Melanoma | Arm 2/ TNBC | Total
Number analyzed (Participants) | 20 | 44 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] — Subject age at time of screening.
  years
    Demographics Across Arms | 62.1 (8.54) | 51.0 (13.37) | 54.4 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex/Gender reported by subject at screening.
  Participants
    Demographics Across Arms: Female | 4 | 43 | 47
    Demographics Across Arms: Male | 16 | 1 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity reported by subject at screening.
  Participants
    Hispanic or Latino | 1 | 6 | 7
    Not Hispanic or Latino | 18 | 37 | 55
    Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race as reported by subject at screening.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 5 | 5
    White | 20 | 37 | 57
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 44 | 64

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint Was ORR, Defined as the Proportion of Subjects Demonstrating CR or PR Based on RECIST v1.1 Criteria.
Description: The best response was defined as the best response recorded from the start of study treatment until the first PD based on RECIST v1.1 or start of new cancer therapy, whichever occurred earlier.
  Response assessment occurred every 6 weeks after the first dose of study drug.
Time Frame: From the start of study treatment until the first PD based on RECIST v1.1 or start of new cancer therapy, whichever occurred earlier, up to 24 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma | Triple Negative Breast Cancer
Number analyzed (Participants) | 20 | 44
Participants
  Complete Response | 1 | 1
  Partial Response | 0 | 5
  Stable Disease | 8 | 17
  Confirmed Progressive Disease | 10 | 19
  Not Evaluable | 1 | 2

2. Secondary Outcome: Time to Response (TTR) Using RECIST v1.1 Criteria
Description: For the subset of subjects with a confirmed CR or PR (RECIST v1.1), TTR was defined as time from the date of the first dose to the first response (the CR/PR prior to the confirmation).
Time Frame: TTR was defined as time from the date of the first dose to the first response, up to 24 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Melanoma | Triple Negative Breast Cancer
Number analyzed (Participants) | 1 | 6
months | 9.66 [9.66 to 9.66] | 2.86 [1.25 to 5.39]

3. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete response rate (CRR) using RECIST v1.1 criteria
Time Frame: The time from the date of the first dose to the first response (CR), up to 24 months.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Melanoma: I4 mg/kg Imprime PGG + 200 mg IV every 3 weeks (Q3W) pembrolizumab in subjects with advanced melanoma
  Pembrolizumab: Pembrolizumab is a humanized monoclonal antibody against the programmed death receptor-1 protein. Pembrolizumab will be given at a fixed dose of 200 mg IV over 30 minutes on Day 1 of each 3-week treatment cycle after the Imprime infusion.
Arm/Group | Melanoma | Triple Negative Breast Cancer
Number analyzed (Participants) | 20 | 44
percentage of patients | 5.3 [0.1 to 26.0] | 2.4 [0.1 to 12.6]

4. Secondary Outcome: Duration of Overall Response (DoR) Using RECIST v1.1 Criteria
Description: For the subset of subjects with a confirmed CR or PR (RECIST v1.1), DoR was defined as the time from the first documented evidence of CR or PR (the response prior to the confirmation) until the time of documented PD (based on radiological assessments per RECIST v1.1) or death due to any cause, whichever occurred earlier.
Time Frame: time from the first documented evidence of CR or PR (the response prior to the confirmation) until the time of documented PD (based on radiological assessments per RECIST v1.1) or death due to any cause, whichever occurred earlier.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Melanoma | Triple Negative Breast Cancer
Number analyzed (Participants) | 1 | 6
Months | 12.68 | 15.24 [4.11 to 20.96]

5. Secondary Outcome: Progression-Free Survival (PFS) Per RECISTv1.1
Description: Progression free survival was defined as the time from the date of the first dose until the first PD or death due to any cause, whichever occurred first.
Time Frame: time from the date of the first dose until the first PD or death due to any cause, whichever occurred first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Melanoma | Triple Negative Breast Cancer
Number analyzed (Participants) | 20 | 44
Months | 1.76 [1.31 to 2.79] | 2.35 [1.35 to 3.98]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of the first dose until the date of death due to any causes.
Time Frame: Time from date of study day 1 until date of death due to any cause.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Melanoma | Triple Negative Breast Cancer
Number analyzed (Participants) | 20 | 44
Months | 8.80 [3.61 to 15.67] | 16.36 [11.10 to 19.22]

7. Other Pre Specified Outcome: Progression Free Survival Based on irRECIST
Description: as for outcome 5
Time Frame: time from the date of the first dose until the first PD or death due to any cause, whichever occurred first.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Melanoma | Triple Negative Breast Cancer
Number analyzed (Participants) | 20 | 44
months | 1.76 [1.31 to 2.99] | 2.86 [1.81 to 4.11]

8. Other Pre Specified Outcome: ORR Based on irRECIST
Description: The best response based on irRECIST was the best response recorded from the start of study treatment until PD (PD per RECIST v1.1 or PD confirmed by irRECIST, whichever was later) or start of new anticancer therapy, whichever occurred earlier.
Time Frame: the best response recorded from the start of study treatment until PD (PD per RECIST v1.1 or PD confirmed by irRECIST, whichever was later) or start of new anticancer therapy, whichever occurred earlier; up to 24 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma | Triple Negative Breast Cancer
Number analyzed (Participants) | 20 | 44
Participants
  Complete Response | 1 | 1
  Partial Response | 0 | 6
  Stable Disease | 8 | 17
  Confirmed Progressive Disease | 2 | 0
  Unconfirmed Progressive Disease | 8 | 18
  Not Evaluable | 1 | 2

9. Post Hoc Outcome: Summary of Overall Response Rate in Subgroup of TNBC Subjects Who Had Received Prior Hormone Therapy
Description: proportion of subjects demonstrating complete response (CR) or partial response (PR) based on RECIST v1.1 thru end of study
Time Frame: The time from the date of the first dose to the first response (CR), up to 24 months.
Population: Evaluable subjects who received prior hormone therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Triple Negative Breast Cancer
Number analyzed (Participants) | 11
Participants | 5

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days post last dose of study drug, up to 25 months.
Arm/Group | Melanoma | Triple Negative Breast Cancer
All-Cause Mortality (participants affected / at risk) | 1/20 | 2/44
Serious Adverse Events (participants affected / at risk) | 3/20 | 9/44
Other Adverse Events (participants affected / at risk) | 20/20 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melanoma (N=20) | Triple Negative Breast Cancer (N=44)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion Related Reactions (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Candida Infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mental status change (Psychiatric disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Melanoma (N=20) | Triple Negative Breast Cancer (N=44)
Fatigue (General disorders) | 11 | 14
Chills (General disorders) | 4 | 13
Axillary pain (General disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 8 | 20
Abdominal pain (Gastrointestinal disorders) | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 3 | 10
Vomiting (Gastrointestinal disorders) | 3 | 12
Diarrhoea (Gastrointestinal disorders) | 2 | 13
Dry Mouth (Gastrointestinal disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 10
Blood bilirubin increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 8
Blood alkaline phosphatase increased (Investigations) | 2 | 4
Dizziness (Nervous system disorders) | 2 | 5
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 9
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 10
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Insomnia (Psychiatric disorders) | 2 | 4
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hypotension (Vascular disorders) | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Pyrexia (General disorders) | 0 | 13
Chest discomfort (General disorders) | 0 | 4
Oedema peripheral (General disorders) | 0 | 4
Pain (General disorders) | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Headache (Nervous system disorders) | 0 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 6
Urinary tract infection (Infections and infestations) | 0 | 4
Pneumonia (Infections and infestations) | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hot flush (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 3
Vision blurred (Eye disorders) | 0 | 4
Tachycardia (Cardiac disorders) | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 3
Hypothyroidism (Endocrine disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT02981303/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT02981303/SAP_001.pdf